CLINICAL TRIAL: NCT03971890
Title: Effectiveness of a Exercise Program Based on Dance Therapy in Fibromyalgia: A Randomized Controlled Trial.
Brief Title: Effectiveness of Dance Therapy in Fibromyalgia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Encarnación Aguilar Ferrandiz, Research and teaching staff of the University of Granada, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ExerFib
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Fibromyalgia
Keywords: Balance; Pain; TUG; Dance
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Dance Therapy; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DanceTherapy Group (Experimental): The experimental group will receive a dance treatment.
  Interventions: Other: Dance therapy
- Control Group (Experimental): The control group will be subjected to a educational treatment.
  Interventions: Other: Educational group

INTERVENTIONS:
Other: Dance therapy — The experimental group will receive a dance treatment.This protocol will be administered at weekly sessions of 60 minutes with a period of 2 times / week with a total of 16 sessions, distributed over a 8-week period. They will be evaluated at baseline, after the end of the last treatment session.
  Other Names: Exercise treatment
  Arms: DanceTherapy Group
Other: Educational group — The control group will receive an educational intervention. They will be evaluated at baseline, after the end of the last treatment session.
  Other Names: Control group
  Arms: Control Group

SUMMARY:
The purpose of this study is to analyze the effects of an intervention with dance on balance,movility, pain and sleep in patients with Fibromyalgia in comparison to a control group that will have an educational intervention.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic disease consisting of widespread pain, fatigue, sleep disturbances, and cognitive impairments, among other symptoms, which affect daily physical activity.

The regular physical exercise improves the functional, physiological, and behavioral components of physical fitness. Dance therapy seems to increase motivation and adherence to therapy, and can provide a real alternative to conventional exercise

The experimental group will receive a dance program treatment .

The control group will receive an educational intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age until 64.
* Being diagnosed with FMS in accordance with American College of Rheumatology - ACR

Exclusion Criteria:

* Participants with diagnoses of other inflammatory rheumatic diseases, previous neurological or orthopedic diseases,
* Use aids for balance, hearing and visual problems.
* Cognitive impairment.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2019-09-21 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | 8 weeks
  Change from de baseline in functional mobility and predict risk of falls. The single-task subscale consists of a measurement of the time in seconds for the patient to rise from sitting in a standard arm chair, walk 3 meters, turn, walk back to the chair, and sit down. The dual task subscale adds a cognitive task (TUGCognitive) or a manual task (TUGManual) to the simple task.

SECONDARY OUTCOMES:
One leg stance | 8 weeks
  Change from de baseline in postural steadiness (static balance) in a static position by registering the number of seconds a person can maintain this position.
SLUMP Test | 8 weeks
  Change from de baseline in the movement of the pain-sensitive nerve structures.
Straight Leg Raise test (SLR) | 8 weeks
  Change from de baseline in the movement of the pain-sensitive nerve structures.
Revised Fibromyalgia Impact Questionnaire (FIQR) | 8 weeks
  Change from the baseline on the impact of symptoms on quality of life in people with fibromyalgia. Questionnaire with 21-items on a visual analogue scale.
Sheehan Disability Scale (SDS) | 8 weeks
  Change from the baseline on the severity of general disability in the items of work, family life/home responsibilities and social life/leisure activities.
Pittsburgh Sleep Quality Index (PSQI) | 8 weeks
  change from the baseline on sleep quality. The self-rated items of the PSQI generate seven component scores (with subscales ranged 0-3): sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping medication, and daytime dysfunction.
Athens Insomnia Scale (AIS) | 8 weeks
  Change from the baseline on insomnia. It is a self-rating instrument of eigth items.
Spanish version of the Brief Pain Inventory questionnaire (CBD) | 8 weeks
  Change from the baseline on the intensity of pain and its impact on activities of daily living.
Health Assessment Questionnaire - Disability Index (HAQ-DI) | 8 weeks
  Change from the baseline on physical disability related to activities of eight categories of daily living over the last week.
Epworth Sleepiness Scale, (EES) | 8 weeks
  Change from thebaseline of the subject's general level of daytime sleepiness.
Minibestest | 8 Weeks
  Change from baseline in Dynamic Balance: areas are anticipatory postural adjustments, reactive postural responses, sensory orientation, and stability in gait. This tool has 14 items, with a maximum score of 28 points.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain